CLINICAL TRIAL: NCT02061904
Title: Prospective Exploratory Study:Bone Mineral Density Changes of the Acetabulum After Revision Hip Arthroplasty Using Bone Impaction Grafting
Brief Title: Bone Mineral Density Changes of the Acetabulum After Revision Hip Arthroplasty Using Bone Impaction Grafting
Acronym: BMD&BIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Job van Susante, MD, PhD, Rijnstate Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BMD&BIG
Record Dates: First submitted 2014-02-09; First posted 2014-02-13 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Disorder of Bone Density and Structure, Unspecified; Satisfaction
MeSH Terms: conditions — Personal Satisfaction | interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Bone Mineral Density (Other): Bone mineral density measurement with "intervention" DEXA at the bone impaction graft site:
  DEXA: dual energy X-ray absorptiometry
  Interventions: Radiation: DEXA: dual energy X-ray absorptiometry
- Hip function (Other): Hip Function/mobility development:
  Harris Hip Score
  Interventions: Other: Harris Hip Score
- pain experience (Other): Pain experiences after surgery in the hip joint VAS-pain
  Interventions: Other: VAS-pain
- General Patients Health condition (Other): Patients health condition monitoring: intervention SF12:
  Short Form Health Survey 12
  Interventions: Other: Short Form Health Survey 12
- Intervention Satisfaction (Other): Patients satisfaction development after the intervention VAS-satisfaction
  Interventions: Other: VAS-satisfaction

INTERVENTIONS:
Radiation: DEXA: dual energy X-ray absorptiometry — Bone mineral density development measured with dual energy X-ray absorptiometry
  Other Names: Bone Mineral Density measurement
  Arms: Bone Mineral Density
Other: Short Form Health Survey 12 — questionnaire for general health monitoring
  Other Names: SF12
  Arms: General Patients Health condition
Other: VAS-satisfaction — questionnaire for intervention satisfaction monitoring
  Other Names: Visual analoge Scale for satisfaction.
  Arms: Intervention Satisfaction
Other: VAS-pain — questionnaire for pain monitoring
  Other Names: visual analog scale for pain
  Arms: pain experience
Other: Harris Hip Score — questionnaire for hip function monitoring
  Other Names: HHS
  Arms: Hip function

SUMMARY:
Prospective explorative study for the investigation of short-term and medium-term outcomes regarding bone mineral density changes after revision hip arthroplasty making use of bone impaction grafting. Outcome measurements will include objective and subjective clinical data, complications and adverse events, radiographic data measurements recorded at several postoperative intervals.

DETAILED DESCRIPTION:
Hypothesis, open questions and specific aims of the project:

We believe that it is important to gain further insight in the process of bone graft remodeling and the preservation of bone stock after bone impaction grafting.

Radiographs are far from conclusive and CT scan can not be repeated on regular intervals for obvious reasons. Prospective follow-up of the BMD of the bone impaction area will contribute to our further understanding. There is no literature available on BMD changes in the acetabulum after bone impaction grafting.

From our recent experiences with earlier research on BMD in specific ROI in the femoral neck we are motivated to further explore the potential of our DEXA technology and software in the field revision hip arthroplasty.

We hypothesize that BMD changes in the bone impaction grafted acetabulum can be adequately monitored with modern DEXA techniques.

Research Questions are:

1. Will bone impaction grafting of the acetabulum result in a well preserved/remodelled bone stock within 2 years after revision hip arthroplasty?
2. Can changes in BMD be interpreted as representative for the process of bone remodelling in the bone impacted area?

   Study design

   This trial as described in this protocol is a prospective explorative follow-up study recording the clinical, radiographic data, and bone mineral density data at specific time intervals (preoperative, within 2 weeks postoperative, at 3months, 6months, 1 year and 2 years postoperative). The data will be collected using SPSS (version 20.)

   Main objective:

   To prospectively assess the BMD at short and medium time intervals in specific ROI as an indicator for the process of bone remodelling and ossification of the bone impaction graft after revision hip arthroplasty..

   Secondary Objectives:

   Clinical scores (SF-12, Oxford Hip score, VAS pain and VAS satisfaction) will be obtained. Vigilant identification of Adverse Events (AEs) will be maintained throughout the study. Mean changes in clinical scores, over time, will also be tested with repeated measurement statistics. Because clinical success is not always indicative of radiographic success and vice versa, correlations will be made.

   Sample size:

   Our study concerns an explorative study in twenty patients.

   Study duration:

   The expected duration of the study is approximately 3 years from the commencement of subject enrollment. Subject enrollment is expected to take 1 year. All subjects will be followed for at least two years after surgery until the last subject achieves two-years follow-up.

   Evaluation criteria

   The study is designed to evaluate possible clinical, radiographic and bone densitometry differences changes after revision hip arthroplasty.

   Evaluation criteria at different follow-up intervals.

   A Clinical:
   * the patient's own evaluation according to the Oxford Score, Dutch translation validated
   * the patient's evaluation of his general health with the SF-12 score , license to validated Dutch translation11
   * the patient's degree of pain and satisfaction with the prosthesis and the procedure.

   B Radiological:
   * X-ray evaluations of implant stability, migration, changing of cup or head angles, radiolucent lines, loosening and osteolysis. X-Rays should preferably be digital, at preoperative, 6 months, 1 year and 2 years.

   C. DEXA bone density measurements

   - Bone density measurements will be performed preoperative on the acetabulum on several regions of interests (ROI's) including the bone impaction grafting area. Once this ROI's of the acetabulum has been determined it can be digitalized and saved into the software, subsequently this ROI can be transported 4 days postoperative and at 4 days postoperative, 6 months, 1 year and 2 years.

   - This method has been tested in our earlier resurfacing study and has proved to be reliable and reproducable.

   - An independent radiologist will do the measurements on the DEXA-scan

   D Survival after revision hip arthroplasty with bone impaction grafting - According to Kaplan Meiers survival rates.

   E Complications and adverse events

   - Early and late complications possibly associated with revision hip arthroplasty and possible relationship with bone impaction grafting and surgical technique.

ELIGIBILITY:
Inclusion Criteria:

1. revision hip arthroplasty with acetabular defects eligible for bone impaction grafting
2. Diagnosis: acetabular osteolytic defects after primary total hip arthroplasty, planned for revision hip arthroplasty with bone impaction grafting.
3. Patient is between 35 and 75 years old.
4. Patient is expected to recover completely.
5. Patient is willing and able to come to follow-up examinations.
6. Patient has signed an informed consent.

Exclusion Criteria:

1. Infection of the hip joint or distant infection (may cause hematogenous spread to the implant site)
2. Hip fractures
3. Patient is younger than 35 years or older than 75 years.
4. Patient is not willing and/or able to come to follow-up examinations
5. Patient has not signed an informed consent
6. Pregnancy

Relative contra-indications:

With regard to the patient's general health:

1. Metabolic disorders or medication (e.g. steroids) which may impair bone formation
2. Osteomalacia
3. Disorders of the immune system, caused by disease or immunosuppressive medication which increase the risk of infection.
4. Poor prognosis for good wound healing: decubitus ulcer, end-stage diabetes, severe protein deficiency and/or malnutrition

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Bone mineral density changes | 24 months
  Acetabular bone mineral density measurements after bone impaction grafting using DEXA, changes in density compared to baseline levels: at < 2weeks postoperative, at 3, 6, 12 and 24 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: J v Susante, MD. PhD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

REFERENCES:
- [Background] Smolders JM, Pakvis DF, Hendrickx BW, Verdonschot N, van Susante JL. Periacetabular bone mineral density changes after resurfacing hip arthroplasty versus conventional total hip arthroplasty. A randomized controlled DEXA study. J Arthroplasty. 2013 Aug;28(7):1177-84. doi: 10.1016/j.arth.2012.08.025. Epub 2012 Dec 6. PMID 23219623
- [Background] Smolders JM, Hol A, Rijnders T, van Susante JL. Changes in bone mineral density in the proximal femur after hip resurfacing and uncemented total hip replacement: A prospective randomised controlled study. J Bone Joint Surg Br. 2010 Nov;92(11):1509-14. doi: 10.1302/0301-620X.92B11.24785. PMID 21037344